CLINICAL TRIAL: NCT03687658
Title: Applying Novel Technologies and Methods to Inform the Ontology of Self-Regulation: Aim 4
Brief Title: Applying Novel Technologies and Methods to Self-Regulation: Behavior Change Tools for Smoking and Binge Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Russell Alan Poldrack, Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 47143; 4UH3DA041713-04 (NIH)
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-08

CONDITIONS: Smoking; Binge Eating; Behavior
MeSH Terms: conditions — Smoking; Bulimia; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binge Eating Group (Experimental): All participants in the study will be invited to use Laddr, described in the intervention section.
  Interventions: Behavioral: Laddr
- Smoking Group (Experimental): All participants in the study will be invited to use Laddr, described in the intervention section.
  Interventions: Behavioral: Laddr

INTERVENTIONS:
Behavioral: Laddr — Laddr is an integrated, personalized, web-based self-regulation assessment and behavior change system. It integrates tools that have been shown to be effective for a wide array of behavioral phenomena ranging from substance use and abuse, mental health, risk-taking, chronic pain management, medication adherence, diet, exercise, diabetes and other chronic disease management, and smoking. The organizational structure, functionality and content within Laddr's system centrally embrace these fundamental aspects of behavior change; thus, the Laddr platform is not "diagnosis-specific" but rather enables integrated care for any combination of individuals' goals, needs, and preferences.

SUMMARY:
This study will evaluate the extent to which we can engage and manipulate putative targets within the self-regulation domain within and outside of laboratory settings in samples of smokers and overweight/obese individuals with binge eating disorder. This is the fourth phase of a study that aims to identify putative mechanisms of behavior change to develop an overarching "ontology" of self-regulatory processes.

ELIGIBILITY:
Inclusion Criteria:

* Understand English sufficiently to provide informed consent
* Right-handed
* Normal or corrected-to-normal vision and no color blindness
* Interest in engaging with Laddr to modify self-regulatory behavior

Additional Inclusion Criteria for Smoking sample:

* Smoke 5 or more tobacco cigarettes/day for past year
* BMI greater than or equal to 17 and less than 27

Additional Inclusion Criteria for Binge Eating Sample:

* BMI greater than or equal to 27 and less than 45
* Weight limit of 350 lbs
* Non-smoking (defined as no cigarettes in past 12 months-this includes former and never smokers)

Exclusion Criteria:

* Significant medical illness
* History of mental disorder due to a medical condition
* Lifetime history of major psychotic disorders (including schizophrenia and bipolar disorder)
* Current use of any medication for psychiatric reasons (including stimulants and mood stabilizers)

Additional Exclusion criteria for Binge Eating Sample:

* Lost weight in recent past (>10 pounds in past 6 months)
* Currently in a weight-loss program (e.g., Weight Watchers, Jenny Craig)
* Currently on a special diet for a serious health condition
* Current engagement in psychotherapy for binge eating disorder

Additional Exclusion Criteria for Smoking Sample:

* Binge eating behavior
* Current engagement in psychotherapy for smoking behavior

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell A Poldrack, PhD, Principal Investigator — Stanford University; Patrick G Bissett, PhD, Study Director — Stanford University
Locations (1):
- Stanford Center for Cognitive and Neurobiological Imaging, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, a de-identified dataset (i.e., stripped of all codes or other information that could be linked back to an individual participant) will be generated and made available to the research community as a whole.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available upon submission of the paper detailing the findings of the research.
Access Criteria: All data will be shared openly, with no restrictions on access.

REFERENCES:
- See also: Related Info — https://scienceofbehaviorchange.org/what-is-sobc/

RESULTS

PARTICIPANT FLOW:
Groups:
- Binge Eating Group: Overweight participants with binge eating disorder were administered Laddr over 4 weeks.
- Smoking Group: Participants who smoked 5 cigarettes or more per day were administered Laddr over 4 weeks.
Period: Overall Study
Arm/Group | Binge Eating Group | Smoking Group
Started | 67 | 24
Completed 1st Scan | 52 | 20
Completed 2nd Scan | 46 | 10
Completed | 46 | 10
Not Completed | 21 | 14

BASELINE CHARACTERISTICS:
Population: Participants who completed both scans are included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Binge Eating Group | Smoking Group | Total
Number analyzed (Participants) | 46 | 10 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.80 (8.27) | 39.7 (8.6) | 34.04 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 2 | 38
  Male | 10 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 1 | 14
  Not Hispanic or Latino | 33 | 9 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 2 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 25 | 7 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46 | 10 | 56

OUTCOME MEASURES:

1. Primary Outcome: Binge Eating Episodes - Loss of Control
Description: Self-reported binge eating episodes is assessed four times daily (morning, early afternoon, late afternoon/evening, and night). A binge eating episode is defined as self-reported overeating and loss of control. Loss of control is assessed by the question "When you ate most recently, did you lose control over your eating?" and is scored as 0 (No), 1 (Yes). Responses provided were averaged across the 28-day period.
Time Frame: 28 days
Population: Participants in the Binge Eating Group only and completed both scans were evaluated for this outcome.
Measure: Mean (Standard Error); unit: episodes
Arm/Group | Binge Eating Group
Number analyzed (Participants) | 46
episodes | 0.212 (0.0213)
Statistical Analysis 1: Comparison: Binge Eating Group; Test type: Other — Generalized linear mixed model (GLMM) with a binomial distribution using a logit link function; p = 0.066, Generalized linear mixed model

2. Primary Outcome: Binge Eating Episodes - Overeating
Description: Self-reported binge eating episodes is assessed four times daily (morning, early afternoon, late afternoon/evening, and night). A binge eating episode is defined as self-reported overeating and loss of control. Overeating is assessed by the question "Since the last prompt, when you ate most recently, did you overeat?" and is scored as 0 (no) or 1 (yes). Responses provided were averaged across the 28-day period.
Time Frame: 28 days
Population: Participants in the Binge Eating Group only and completed both scans were evaluated for this outcome.
Measure: Mean (Standard Error); unit: episodes
Arm/Group | Binge Eating Group
Number analyzed (Participants) | 46
episodes | 0.286 (0.0235)
Statistical Analysis 1: Comparison: Binge Eating Group; Test type: Other — Generalized linear mixed model (GLMM) with a binomial distribution using a logit link function; p = 0.273, Generalized linear mixed model

3. Primary Outcome: Number of Cigarettes Smoked Per Day
Description: Self-reported smoking assessed four times daily (morning, early afternoon, late afternoon/evening, and night). A smoking episode is defined as self-reported smoking of more than zero cigarettes and is assessed by the question "Since the last prompt, how many cigarettes have you smoked?" Participants are asked to input a number into a number field and this was averaged over the 28 day period.
Time Frame: 28 days
Population: Participants in the Smoking Group only and completed both scans were evaluated for this outcome.
Measure: Mean (Standard Error); unit: cigarettes per day
Arm/Group | Smoking Group
Number analyzed (Participants) | 10
cigarettes per day | 2.97 (0.547)
Statistical Analysis 1: Comparison: Smoking Group; Test type: Other — Generalized linear mixed model (GLMM) with a Poisson distribution using a log link function; p = 0.403, Generalized linear mixed model

ADVERSE EVENTS:
Time Frame: Average approximately 5 weeks
Arm/Group | Binge Eating Group | Smoking Group
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/24
Other Adverse Events (participants affected / at risk) | 0/67 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT03687658/Prot_001.pdf
  • Statistical Analysis Plan (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT03687658/SAP_002.pdf
  • Informed Consent Form (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT03687658/ICF_000.pdf